CLINICAL TRIAL: NCT03912623
Title: Evaluation of the Benefit at 6 Months of a 3 Weeks Spa Treatment in the Type 2 Diabetic Patient. Multicenter Randomized Therapeutic Trial
Brief Title: Evaluation of the Benefit at 6 Months of a 3 Weeks Spa Treatment in the Type 2 Diabetic Patient.
Acronym: DIABEO2THERMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: TIMC-IMAG (Other); Floralis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A00603-54
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus; Physical Activity; Dietetic Rules; Therapeutic Education
Keywords: HbA1c; Diabetes; Type 2
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Multicenter, Controlled, Randomized, Open Group Therapeutic Trial
Masking Description: We wil use the zelen randomisation to minimize patient disappointment. The patient will be advice of only one group (3 weeks SPA treatment or only a week end access to the SPA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 weeks SPA Treatment (Active Comparator): 3-week thermal cure:
  * Spa treatment harmonized in the different stations
  * Therapeutic education workshops and conferences common to all stations in the form of practical workshops during supervised lunches
  * Adapted physical activity, workshops are common to all spas and use an electric bike suitable for health (VELIS) with briefing and debriefing. An APA (Adapted Physical Activity) coaching consultation at the end of the cure for personalized post-cure programs and objectives is planned as well as a telephone or internet coaching during the 5 months post-cure (objectives and adaptation, motivation)
  * Maintenance of the usual treatment within 6 months post randomization with optimization of the therapeutic target in HbA1c and therapeutic strategies by the software Diascope and / or HAS
  * Information booklet for inclusion (French Association of Diabetics)
  Interventions: Other: SPA Treatment with therapeutic education and physical activity
- Discovery week end (Sham Comparator): Maintenance of usual treatment within 6 months post-randomization with optimization of the therapeutic target in HbA1c and therapeutic strategies by Diascope and HAS software In addition, a "discovery" access to the baths of 2-3 days will be offered to patients. Finally, the information booklet on diabetes will be given at the inclusion (French Federation of Diabetics).
  Interventions: Other: Week end

INTERVENTIONS:
Other: SPA Treatment with therapeutic education and physical activity — 3 weeks SPA Treatment plus therapeutic education plus physical activity
  Arms: 3 weeks SPA Treatment
Other: Week end — access to the station for a week end after maintenance of usual treatment during 6 months
  Arms: Discovery week end

SUMMARY:
Diabetes mellitus is a metabolic disorder characterized by chronic hyperglycemia due to deficiency in either insulin secretion, insulin action, or both. There are different types of diabetes. The most common nowadays is type 2 diabetes, characterized by insulin resistance and a relative deficiency of insulin secretion, either of which may dominate to a varying degree. This form of diabetes occurs mainly in mature adults but can also occur at a younger age, or even during adolescence.

According to estimates, the number of diabetic subjects in the world increased from 153 million in 1980 to 347 million in 2008. In France, the prevalence of diabetes treated increased from 2.6% to 4.4% between 2000 and 2009, reaching nearly 3 million people. Type 2 diabetes accounts for 92% of cases of diabetes treated, and its share continues to increase due to a relative stability of type 1 diabetes and a steady increase in type 2 diabetes (5.4% per year). The aging of the population, the increase in obesity and the lack of physical activity contribute to the development of type 2 diabetes. According to the Entred study conducted in France between 2001 and 2007, four out of five type 2 diabetic patients were either overweight (39%) or obese (41%).

In the long term, unbalanced diabetes exposes to macro-vascular complications such as myocardial infarction and stroke, and microvascular complications affecting the peripheral nervous system, kidneys, retina may result in amputation of the lower limb, renal failure and blindness, respectively. As a result, the risk of death for diabetics is at least twice as high as for non-diabetics.

However, a good control of the disease by a lifestyle adaptation (lifestyle and dietary measures, physical activity) with good medical care, and possibly pharmacological, can avoid or significantly reduce the risk of complications. The purpose of dietary and lifestyle measures is to reduce hyperglycaemia and to control the weight of the patient. The implementation of effective dietary measures is a necessary prerequisite for the medication treatment of glycemic control and their application should be continued throughout the course of treatment. The treatment of other cardiovascular risk factors and complications of diabetes is also essential for the management of the diabetic patient.

The HAS (Haute Autorité de Santé : High Authority of Health) in its latest recommendations for a drug strategy for glycemic control of type 2 diabetes emphasizes that the short-term goal of decreasing hyperglycemia is the improvement of symptoms (thirst, polyuria, asthenia, weight loss and fuzziness visual) and the prevention of acute complications (infectious and hyperosmolar coma). The longer-term goal is the prevention of chronic microvascular complications (retinopathy, nephropathy and neuropathy), macrovascular (myocardial infarction, stroke, and peripheral arterial occlusive disease) and decreased mortality. The HAS notes, however, that HbA1c as a criterion for substituting morbidity and mortality endpoints in type 2 diabetes is not sufficiently supported in the scientific literature.

Be that as it may, HAS recommends individualizing the goal of glycemic control according to the profile of the patient and in particular to mobilize the recommended therapeutic means to reach the HbA1c target, in particular the dietary and hygiene measures. The data in the literature do not allow to define a lower limit for the HbA1c target. For most type 2 diabetic patients, an HbA1c target of less than or equal to 7% is recommended.

A target of 6.5% is recommended for newly diagnosed patients with no history of cardiovascular disease and a life expectancy of more than 15 years, as well as for women during pregnancy. An HbA1c target of 8% or less is recommended for patients with proven severe comorbidity and / or limited life expectancy (<5 years), or with advanced or long-lasting macrovascular complications diabetes (> 10 years) and for whom the target of 7% is difficult to achieve because drug intensification causes severe hypoglycaemia, or with a history of macrovascular complication considered as advanced, or with severe chronic renal insufficiency or (stages 4 and 5), as well as for the so-called frail elderly. For elderly people who are "sick", the priority is to avoid acute complications due to diabetes (dehydration, hyperosmolar coma) and hypoglycaemia; Pre-meal capillary glucose values of between 1 and 2 g / l and / or an HbA1c level of less than 9% are recommended. There are many molecules available on the pharmaceutical market to treat this disease (biguanides, hypoglycemic sulfonamides, DPP-4 inhibitors, GLP-1 analogues, alpha-glucosidase inhibitors, insulin, etc.). It is important to choose, depending on the clinical profile of the patient, the molecule (s) to be combined in order to achieve the glycated hemoglobin targets set by health organizations.

DETAILED DESCRIPTION:
In recent years, many medical decision support software (diagnostic or therapeutic) have emerged to help doctors in their choices. For type 2 diabetes, apart from a decision-making aid tool posted on the HAS website, the Diascope tool can be cited. A group of 12 European experts came together to create this software to help doctors when diabetic patients do not reach their goal. They worked on more than 2000 clinical scenarios and thus established therapeutic recommendations. They prioritized the recommendations in 3 levels. For each patient profile, the most appropriate therapeutic proposals appear in green, inappropriate options appear in red, and acceptable but uncertain options appear in yellow.

These two tools can help optimize patient management by finding the therapeutic strategy that is closest to the recommendations that are adapted to each patient.

Therapeutic education, which has a key role in the care of these patients, has a demonstrated impact on quality improvement. In this prospective study, the authors also found a link between improved quality of life and lower HbA1c. This study uses the Diabetes Quality of Life (DQOL) score. A more appropriate score allowing a customization of the elements constituting the quality of life is the Audit of Diabetes-Dependent Quality of Life score (ADDQOL score).

Physical activity is recommended for multiple reasons in Health. The summary of Inserm's collective expertise perfectly summarizes the benefits and the modalities of a physical activity for Health.

There are clear international recommendations on the subject of moderate physical activity of at least 150 minutes per week, for example on the World Health Organization website or in the text of the recommendations of the American College of Sport Medicine and the American Heart Association. Adaptations of these recommendations for older people are also available. Walking and cycling are the two physical activities most cited in these documents because of their progressive and mild characteristics particularly suitable for patients with rheumatological indications and / or significant overweight. However, the practice of cycling can, depending on the natural terrain, involve efforts and pressures in joints and musculotendinous too important.

This will often be the case in the natural environment of the most often hilly spas. In addition, there are many practical or psychological obstacles to cycling in a population of patients suffering from chronic pathologies: "it's too hard", "I do not know how to do it anymore", "it's for young people "," I am less strong than the others so I can not accompany them in their outings ".... The electric assistance bicycle (EVA) can then be useful. A very comprehensive report from the DGS (Direction Générale de la Santé : General Health Direction) of the Canton of Geneva takes stock of the positive impact of the dissemination of routine use of VAE (Available on http://www.impactsante.ch/pdf/EIS_VAE_2006.pdf). Still in Switzerland, J Welker, despite a provocative title, concludes that "The electric-assisted bicycle (EVA) is a physical activity in its own right and represents a means to fight sedentariness". These authors suggest from a study conducted in Lausanne that VAE even with a high attendance represents a real physical activity (> 6 MET) on hilly paths.

It has been shown on small series with real-time measurements of the effort that the VAE with strong attendance was equivalent to a brisk walk and that the VAE with moderate assistance was intermediate in terms of physical effort between brisk walking and cycling without. It has also been shown that the use of VAE can achieve the objectives recommended for the practice of physical activity.

The hydrotherapy has demonstrated its effectiveness especially for indications rheumatology and for the management of obesity (indication metabolic diseases). The benefit of the multifaceted actions implemented during a spa treatment concerns the symptoms, the reduction of pain and / or weight loss. As a result, randomized controlled trials have shown a benefit on quality of life.

Metabolic disorders and especially diabetes and overweight are an indication of thermal cures. Two studies have shown positive results of a thermal cure on metabolic disorders. The first is a multicentre study in overweight or obese subjects (8% of whom are diabetic) who has demonstrated a significant benefit on weight and body mass index (BMI) of a spa treatment and the maintenance of this condition. improvement one year later compared to a control group. The second is a monocentric study in which a disappearance of a metabolic syndrome was observed one year after a spa treatment for 50% of patients included and 76% of patients followed at one year. Finally, an improvement in weight, BMI and fasting blood glucose at the end of a spa treatment was found in a preliminary study in 21 subjects with type 2 diabetes, with a decrease of 0.5% in glycated hemoglobin (HbA1c) 3 months after the beginning of the treatment.

These positive data on parameters strongly correlated with diabetes (weight, BMI, metabolic syndrome), and on the glycemic parameters of a preliminary study with a small number of diabetic patients justify the completion of a multicenter study to evaluate the benefit to a patient. year of a 3 weeks spa treatment in the type 2 diabetic patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with type 2 diabetes defined by (HAS 2013):

   * a blood glucose level above 1.26 g / l (7.0 mmol / l) after an 8-hour fast and checked twice;
   * or the presence of symptoms of diabetes (polyuria, polydipsia, weight loss) associated with blood glucose (on venous plasma) greater than or equal to 2 g / l (11.1 mmol / l);
   * or blood glucose (on venous plasma) greater than or equal to 2 g / l (11.1 mmol / l) 2 hours after an oral load of 75 g of glucose (criteria proposed by the World Health Organization).
2. Patient with HbA1c at inclusion> 7 and <12% (on an HbA1c dose less than 6 months old at the prescreening)
3. Patient with a BMI ≥ 25 and a weight ≤ 125 kg
4. Patient with appropriate treatment
5. Age ≥ 18 years
6. Available to go on treatment in 6 weeks after inclusion
7. Available for a 12-month follow-up
8. Affiliated to the social security or beneficiary of such a scheme

Exclusion Criteria:

1. Diabetes type 1 or secondary
2. Patient with GFR (glomerular filtration rate) <50 ml / min (MDRD formulation) for at least 1 year.
3. Unstable diabetes defined by the knowledge of the questioning of a change in HbA1c of +/- 1 in the last 6 months.
4. With known serious comorbidity and / or limited life expectancy (<5 years), or with advanced macrovascular complications: in particular cardiovascular (acute coronary diseases and / or stroke in the last 6 months) and renal
5. Severe psychiatric pathology or psychosis
6. Pregnant woman, parturient or breastfeeding
7. Contraindication to hydrotherapy
8. Patient with a contraindication to moderate physical activity or cycling (acute coronary artery disease less than 2 years old, musculoskeletal problem of the spine or lower limbs incompatible with cycling).
9. No previous spa treatment for "Digestive disorders and metabolic diseases" in the current the spa year.
10. Person deprived of liberty or legal protection measure
11. Subject participating to an other clinical study interventional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c evolution | 6 months
  Difference in mean HbA1c between the intervention group (spa treatment) at 6 months post start of treatment and the reference group (usual care) at 6 months post randomization taking into account (Ancova) the last value of d HbA1c available (at baseline or at baseline).

SECONDARY OUTCOMES:
Qualitative evolution of HbA1c | 6 months
  Success defined by three criteria for the evolution of HbA1c: percentage of patients with HbA1c less than or equal to 7% (HAS Criterion) or percentage of patients with at least 1% reduction in HbA1c or percentage of patients who achieved the target HbA1c defined at inclusion
Quantitative evolution of HbA1c | 12 months
  HbA1C at 12 months in quantitative value adjusted to the value at inclusion
Evaluation of the specific quality of life: (ADDQOL) | 6 and 12 months
  The ADDQOL (Audit of Diabetes-Dependent Quality of Life Scale) contain 19 domains.
  These 19 domains ask the respondents to evaluate how their life would be if they did not have diabetes. The scales range from -3 to +1 for 19 life domains (impact rating) and from 0 to +3 in attributed importance (importance rating). A weighted score for each domain is calculated as a multiplier of impact rating and importance rating (ranging from -9 to +3). Lower scores reflect poorer QoL. Finally, a mean weighted impact score (ADDQOL score) is calculated for the entire scale across all applicable domains.
Evaluation of the overall quality of life: (EQ5D- 3L) | 6 and 12 months
  Euroquol 5D (EQ5D- 3L) quality of life scale. Euroquol 5D (EQ5D- 3L) quality of life scale. EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ5D-3L contains 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression).
  Each dimension has 3 levels (no problem, some problem, extreme problem).
Medical care assessment | 6 and 12 months
  evaluation of the medical care of patients (treatments, paramedical procedures, hospitalizations ...), comparison between the 2 groups of treatment modifications.
Biological parameters evolution | 6 and 12 months
  Evolution of biological parameters
Overweight evolution BMI | 6 and 12 months
  Evolution of overweight (BMI)
Overweight evolution abdominal perimeter | 6 and 12 months
  Evolution of overweight (abdominal perimeter)
Clinical repercussions evolution | 6 and 12 months
  Evolution at 6 months and 12 months of the clinical repercussions of diabetes (collection of declarative SAEs with validation by a committee). Analysis of hospitalizations related to diabetes (macro and microvascular repercussions, metabolic complications, severe hypoglycaemia).
Physical activity measurement : (GPAQ score) | 6 and 12 months
  Measurement of physical activity at 6 and 12 months with Global Physical Activity Questionnaire (GPAQ score).The Global Questionnaire on Physical Exercise (GPAQ), has 16 questions.
  The score obtained makes it possible to establish three profiles: insufficient level of physical activity, level according to the recommendations, high level
Physical performance measurement | During SPA therapy
  Pre and post cure measurement of physical performance. Evolution of performances during bike rides (VELIS). Profile of the parameters recorded on the VELIS (cardio, speed, electric power supplied by the engine, pressure on the pedals) at the beginning and end of treatment on the same reference course.
Self-esteem (Rosenberg score) assessment | 6 and 12 months
  Assessment of self-esteem building with the Rosenberg score.The Rosenberg score is between 10 and 40.
  The interpretation of the results is identical for a man or a woman. score below 25, self-esteem is very low. score between 25 and 31, self-esteem is low. score between 31 and 34, self-esteem is average. score between 34 and 39, self-esteem is strong. score above 39, self-esteem is very strong
Treatment compliance | 6 months
  Evaluate the participation in thermal treatment, education and physical activity
Therapeutic objectives evaluation | 3 and 6 months
  Evaluation of the achievement of educational objectives of health behaviors by intermediate telephone follow-up.
Side effects evaluation | 6 and 12 months
  Evaluation of the side effects of the thermal treatment (SAE reporting). Evaluation of all adverse events attributable to treatment, or not, according to the usual criteria of pharmacovigilance in clinical trials
Subgroup analysis | 6 months
  Sub group analysis on the primary outcome measure (stratification on primo spa therapy and age (median 62 years)).

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - ROUSSEL Ludivine, Amiens
  - SOUDET Simon, Amiens
  - ODDOU Christel, Annecy
  - CLERGEOT Annie, Besançon
  - WATERLOT, Chambéry
  - DAOUDI, Corbeil-Essonnes
  - PENFORNIS Alfred, Corbeil-Essonnes
  - BETRY Cécile, Grenoble
  - PARADIS Sabrina, Montmélian

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danaei G, Finucane MM, Lu Y, Singh GM, Cowan MJ, Paciorek CJ, Lin JK, Farzadfar F, Khang YH, Stevens GA, Rao M, Ali MK, Riley LM, Robinson CA, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Blood Glucose). National, regional, and global trends in fasting plasma glucose and diabetes prevalence since 1980: systematic analysis of health examination surveys and epidemiological studies with 370 country-years and 2.7 million participants. Lancet. 2011 Jul 2;378(9785):31-40. doi: 10.1016/S0140-6736(11)60679-X. Epub 2011 Jun 24. PMID 21705069
- [Background] Ampudia-Blasco FJ, Benhamou PY, Charpentier G, Consoli A, Diamant M, Gallwitz B, Khunti K, Mathieu C, Ridderstrale M, Seufert J, Tack C, Vilsboll T, Phan TM, Stoevelaar H. A decision support tool for appropriate glucose-lowering therapy in patients with type 2 diabetes. Diabetes Technol Ther. 2015 Mar;17(3):194-202. doi: 10.1089/dia.2014.0260. Epub 2014 Oct 27. PMID 25347226
- [Background] Debaty I, Halimi S, Quesada JL, Baudrant M, Allenet B, Benhamou PY. A prospective study of quality of life in 77 type 1 diabetic patients 12 months after a hospital therapeutic educational programme. Diabetes Metab. 2008 Nov;34(5):507-13. doi: 10.1016/j.diabet.2008.03.007. Epub 2008 Sep 30. PMID 18829362
- [Background] Bradley C, Todd C, Gorton T, Symonds E, Martin A, Plowright R. The development of an individualized questionnaire measure of perceived impact of diabetes on quality of life: the ADDQoL. Qual Life Res. 1999;8(1-2):79-91. doi: 10.1023/a:1026485130100. PMID 10457741
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131
- [Background] Hanh T, Serog P, Fauconnier J, Batailler P, Mercier F, Roques CF, Blin P. One-year effectiveness of a 3-week balneotherapy program for the treatment of overweight or obesity. Evid Based Complement Alternat Med. 2012;2012:150839. doi: 10.1155/2012/150839. Epub 2012 Dec 24. PMID 23346190
- [Background] Gin H, Demeaux JL, Grelaud A, Grolleau A, Droz-Perroteau C, Robinson P, Lassalle R, Abouelfath A, Boisseau M, Toussaint C, Moore N. Observation of the long-term effects of lifestyle intervention during balneotherapy in metabolic syndrome. Therapie. 2013 May-Jun;68(3):163-7. doi: 10.2515/therapie/2013025. Epub 2013 Jul 26. PMID 23886461